CLINICAL TRIAL: NCT00279422
Title: A Phase 2/3, Randomized, Double-blind, Placebo-controlled, Multicenter Study of Visilizumab in Subjects With Intravenous Steroid-Refractory Ulcerative Colitis
Brief Title: A Study of Visilizumab in Subjects With Intravenous Steroid-Refractory Ulcerative Colitis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: DMC recommendation, no efficacy
Sponsor: Facet Biotech (Industry)
Collaborators: PDL BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 291-415
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Ulcerative Colitis
Keywords: Intravenous, Steroid-Refractory, Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — visilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: visilizumab
- visilizumab (Experimental)
  Interventions: Drug: visilizumab

INTERVENTIONS:
Drug: visilizumab
  Arms: visilizumab
Drug: visilizumab
  Arms: placebo

SUMMARY:
The purpose of this study is to compare the efficacy of visilizumab to placebo in subjects with intravenous steroid-refractory ulcerative colitis.

DETAILED DESCRIPTION:
PDL BioPharma, Inc. was formerly known as Protein Design Labs, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age or older.
* Diagnosis of ulcerative colitis (UC) verified by endoscopy within 60 months prior to consent.
* Severe active disease, as defined by a Modified Truelove & Witts Severity Index (MTWSI; also known as Lichtiger score) ≥ 11 at consent, with a confirmatory MTWSI ≥ 10 on or after the fifth consecutive day of intravenous (IV)steroids and within 1 day prior to randomization.
* Mayo score ≥ 10 and Mayo mucosal subscore ≥ 2 after a minimum of 3 consecutive days (ie, on or after the fourth consecutive day) of IV steroids.
* Adequate contraception from the day of consent through 3 months after the last dose of study drug.
* Negative serum pregnancy test.
* Negative Clostridium difficile test.
* Signed and dated informed consent and Health Insurance Portability and Accountability Act (HIPAA) if applicable.

Exclusion Criteria:

* UC requiring immediate intervention or toxic megacolon requiring imminent intervention.
* History of total proctocolectomy, or subtotal colectomy with ileorectal anastomosis.
* Presence of Ileostomy.
* White blood cell count less than 2.5 x 10^3/mcL; platelet count less than 150 x 10^3/mcL; or hemoglobin level less than 8 g/dL.
* Active medically significant infections, particularly those of viral etiology, eg, known cytomegalovirus (CMV) colitis. This includes any incidence of medically significant opportunistic infections within the past 12 months.
* Live vaccination within 6 weeks prior to randomization.
* Significant organ dysfunction, including cardiac, renal, liver, central nervous system (CNS), pulmonary, vascular, gastrointestinal, endocrine, or laboratory abnormality.
* History of myocardial infarction, coronary artery disease, congestive heart failure, or arrythmias within 6 months prior to consent.
* History or treatment of lymphoproliferative disorder (LPD) or malignancy within the past 5 years (excluding nonmelanoma skin cancer or carcinoma in situ of the cervix).
* Seropositivity for infection with human immunodeficiency virus (HIV-1), hepatitis B virus (HBV) surface antigen, or hepatitis C virus (HCV).
* Pregnancy or nursing.
* Treatment with a first dose of infliximab or another anti-tumor necrosis factor (TNF)-α drug within 4 weeks of randomization, or treatment with a subsequent dose of an anti-TNF-α drug within 2 weeks of randomization.
* Treatment with cyclosporine or tacrolimus (FK506) within 2 weeks prior to randomization.
* Treatment with any other investigational drugs or therapies within 60 days prior to randomization, except those mentioned in the two exclusion criteria above.
* Unable or willing to discontinue any UC drug (including, but not limited to 6-mercaptopurine, azathioprine, or methotrexate), except glucocorticoids or 5-ASA, immediately prior to randomization.
* Nontherapeutic levels of chronic antiseizure medications in subjects with a prior history of seizures.
* Any condition that, in the investigator's opinion, makes the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (17):
  - Los Angeles, California
  - San Francisco, California
  - Gainesville, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Rochester, Minnesota
  - New York, New York
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Galveston, Texas
- Australia (9):
  - Camperdown, New South Wales
  - Liverpool, New South Wales
  - Herston, Queensland
  - South Brisbane, Queensland
  - Box Hill, Victoria
  - Bedford Park
  - Fitzroy
  - Fremantle
  - Parkville
- Vienna, Austria
- Belgium (3):
  - Ghent
  - Leuven
  - Roeselare
- Canada (2):
  - Calgary, Alberta
  - London, Ontario
- Czechia (2):
  - Brno
  - Prague
- France (7):
  - Amiens, Cedex
  - Clichy
  - Lille
  - Marseille
  - Nantes
  - Nice
  - Paris
- Germany (8):
  - Berlin
  - Frankfurt
  - Freiburg im Breisgau
  - Hanover
  - Kiel
  - München
  - Rostock
  - Stuttgart
- Hungary (7):
  - Argenti Döme
  - Budapest
  - Csabai Kapu
  - Debrecen
  - Győr, Vasvári Pál
  - Szekszárd
  - Veszprém
- Israel (3):
  - Haifa
  - Tel Aviv
  - Tel Litwinsky
- Netherlands (2):
  - Amsterdam
  - Rotterdam
- Norway (3):
  - Oslo
  - Prinsens
  - Tromsø
- Mickieviczova, Slovakia
- Ukraine (3):
  - Kharkiv
  - Kyiv
  - Odesa

REFERENCES:
- [Derived] Sandborn WJ, Colombel JF, Frankel M, Hommes D, Lowder JN, Mayer L, Plevy S, Stokkers P, Travis S, Van Assche G, Baumgart DC, Targan SR. Anti-CD3 antibody visilizumab is not effective in patients with intravenous corticosteroid-refractory ulcerative colitis. Gut. 2010 Nov;59(11):1485-92. doi: 10.1136/gut.2009.205443. PMID 20947884